CLINICAL TRIAL: NCT06497725
Title: Remote Teleguidance-facilitated Airway Management in Prehospital Emergency Medical Services: A Randomized Controlled Simulation Study
Brief Title: Teleguidance-facilitated Airway Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ibrahim Ulas Ozturan, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GOKAEK-2024/07.13
Record Dates: First submitted 2024-06-28; First posted 2024-07-12 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Telemedicine; Intubation; Difficult or Failed; Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleguidance-facilitated Airway Management (Experimental): The airway expert able to remotely access to videolaryngoscopy monitor will provide verbal feedback during the endotracheal intubation.
  Interventions: Device: Teleguidance-facilitated Airway Management
- Standard Airway Management (No Intervention): Operator will use standard videolaryngoscopy without expert feedback during the endotracheal intubation.

INTERVENTIONS:
Device: Teleguidance-facilitated Airway Management — tele-guidence will be provided by an experienced airway expert
  Arms: Teleguidance-facilitated Airway Management

SUMMARY:
The advent of telemedicine has introduced teleguidance as a promising support to enhance endotracheal intubation skills among inexperienced operators. Several studies showed the effectiveness of supervisor assisted ETI using the various VL devices and commercial videoconferencing softwares. However, recent developments in VL technologies introduced the VL integrated videoconferencing features for this purpose. Scoper VL device (Technomedicare Inc, Turkiye) developed a real-time teleconsultation feature for difficult airway scenarios to be assisted by experts during the procedure. However, the literature is very limited about the effectiveness and feasibility of teleguidance-facilitated airway management.

This high-fidelity simulation study aims to assess impact of teleguidance-facilitated airway management on the success of ETI performed by inexperienced operators in a mobile ambulance.

ELIGIBILITY:
Inclusion Criteria:

* All paramedic students who completed their airway management training

Exclusion Criteria:

* The trainees who did not consent to participate
* The trainees who did not complete the VL training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Rate of first attempt success (n,%) | Measured at the 60-second mark.
  Visualization of the endotracheal tube passing between the vocal cords within the first 60 seconds of the procedure.

SECONDARY OUTCOMES:
Intubation duration (seconds) | procedure (Measured at the confirmation of the tube passed between vocal cords.)
  Duration between the passage of the endotracheal tube through the lips and its pass between the vocal cords
Operator confidence assessed by Likert Scale. | At the end of the procedure
  Self-evaluation of procedure confidence using 7-point Likert Scale
Feasibility of intubation assessed by Likert Scale. | At the end of the procedure
  Self-evaluation of methods feasibility using 7-point Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Ozturan, Study Chair — Kocaeli University
Locations (1):
- Kocaeli University Medical Faculty Emergency Medicine Department, Kocaeli, Turkey (Türkiye)